CLINICAL TRIAL: NCT00504270
Title: A Randomized, Placebo-controlled Dose-ranging Pilot Study to Assess the Effect on Clinical Response, and the Safety and Tolerability of R3421 in Patients With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: A Study of R3421 in Patients With Moderate to Severe Chronic Plaque Psoriasis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NS20454
Record Dates: First submitted 2007-07-18; First posted 2007-07-19 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo (Placebo Comparator): po daily
  Interventions: Drug: Placebo
- RG3421 120mg (Experimental): 120mg po daily
  Interventions: Drug: RG3421 120mg
- RG3421 20mg (Experimental): 20mg po daily
  Interventions: Drug: RG3421 20mg

INTERVENTIONS:
Drug: Placebo — po daily
  Arms: Placebo
Drug: RG3421 120mg — 120mg po daily
  Arms: RG3421 120mg
Drug: RG3421 20mg — 20mg po daily
  Arms: RG3421 20mg

SUMMARY:
This study will investigate the safety, efficacy and pharmacokinetics of R3421 in patients with moderate to severe chronic plaque psoriasis. Patients will be randomized to one of 3 treatment groups to receive once daily oral treatment with a)R3421 20mg, b)R3421 120mg, or c)placebo. The anticipated time on study treatment is <3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-70 years of age;
* medically stable, moderate to severe chronic plaque psoriasis.

Exclusion Criteria:

* any skin condition which may interfere with evaluation of the effect of study medication on plaque lesions;
* confounding or concomitant condition or treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs), laboratory parameters, pharmacokinetics | Throughout study

SECONDARY OUTCOMES:
Change from baseline in static physician global assessment (PGA) score, Psoriasis Area and Severity Index (PASI) and exploratory biomarkers | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (14):
- United States (14):
  - Hot Springs, Arkansas
  - Little Rock, Arkansas
  - Santa Monica, California
  - Alpharetta, Georgia
  - East Windsor, New Jersey
  - Albuquerque, New Mexico
  - New York, New York
  - Stony Brook, New York
  - Winston-Salem, North Carolina
  - Providence, Rhode Island
  - Nashville, Tennessee
  - Galveston, Texas
  - San Antonio, Texas
  - Webster, Texas